CLINICAL TRIAL: NCT03504748
Title: Deep rTMS in Parkinson Disease Pain Syndromes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Daniel Ciampi Araujo de Andrade, MD, PhD, MD, PhD (Head of Pain Division), University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VRBDCA
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Pain; Parkinson Disease
Keywords: deep repetitive transcranial magnetic stimulation; chronic pain; parkinson; treatment; non-motor symptom
MeSH Terms: conditions — Pain; Parkinson Disease; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- deep rTMS-active doble coil (Active Comparator): patients undergoing of deep rTMS real with doble coil
  Interventions: Device: deep rTMS
- deep rTMS-sham (Sham Comparator): patients undergoing to placebo deep rTMS
  Interventions: Device: placebo deep rTMS

INTERVENTIONS:
Device: deep rTMS
  Arms: deep rTMS-active doble coil
Device: placebo deep rTMS
  Arms: deep rTMS-sham

SUMMARY:
Pain is the most prevalent non-motor symptom in Parkinson disease, and the motor improvement not always is related to the pain improvement with the medication treatment. By this, we are testing a non-invasive method called transcranial magnetic stimulation as an alternative to treat pain related to Parkinson disease. This technique can lead to either inhibitory or excitatory effects in brain circuits depending on stimulation parameters, and is known to provide analgesic effects.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson disease
* Signed term of informed consent
* Parkinsson disease related pain

Exclusion Criteria:

* Trauma of Skull, epilepsy don't treated
* Use of medications decrease the seizure threshold
* Patients in use of drugs, how cocaine and alcohol
* neurosurgical clips, pacemakers, increased intracranial pressure (risk of sequelae after seizure)
* Pregnant or lacting women
* Moderate or severe cognitive impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-07-20 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in baseline of Pain | base line (moment of inclusion), day 15th, day 45th and in the last day of the sessions of rTMS (4X in two months)
  assessing by Visual Analog Scale for Pain (VAS). This scale range from 0 (no pain) to 10 (maximum pain), being considered an effective improvement in the patient's pain when the pain decreases at least in 30% from the basal score.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (HC/FMUSP), São Paulo, São Paulo, Brazil